CLINICAL TRIAL: NCT03596229
Title: Incidence of Postoperative Major Adverse Cardiac Events in the Patients Underwent Carotid Endarterectomy: A Single Center Retrospective Study
Brief Title: Major Adverse Cardiac Events After Carotid Endarterectomy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Aphichat Suphathamwit,, Lecturer, Mahidol University
Other Study IDs: 2018_1
Record Dates: First submitted 2018-07-05; First posted 2018-07-23 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Carotid Stenosis; Carotid Endarterectomy; Adverse Cardiac Events
Keywords: carotid endarterectomy; adverse cardiac events
MeSH Terms: conditions — Carotid Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Carotid endarterectomy is the operation for curing the significant carotid artery stenotic patients who are also at high cardiac risk. This retrospective study is to find out the incidence and risk factors related.

DETAILED DESCRIPTION:
The investigator plan to retrospectively investigate 175 carotid endarterectomy patients in Siriraj hospital to find the incidences of major adverse cardiac events, including

* Myocardial infarction is defined as rising of cardiac bio-markers in the setting of myocardial ischemia (Relevant anginal symptoms, ECG changes or Imaging e.g. Echocardiography)2,10
* Significant arrhythmia is defined as symptomatic or causing hemodynamic changes without other explainable causes.
* Heart failure is defined according to Modified Framingham criteria3
* Cardiac death is defined as mortality in association and as a direct result from myocardial infarction, arrhythmia or heart failure

if possible, the investigators will try to find the associate or risk factors for those events.

ELIGIBILITY:
Inclusion Criteria:

* Every patients undergoing carotid endarterectomy in Siriraj hospital

Exclusion Criteria:

* Patients with other simultaneous surgery with carotid endarterectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The carotid stenotic patents scheduled for carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events after carotid endarterectomy | 7 days
  Major adverse cardiac event included myocardial infarction, significant arrhythmia, heart failure and cardiac arrest

SECONDARY OUTCOMES:
associate factors with adverse cardiac event | 7 days
  Analysis of potential factors associated with major adverse cardiac event after carotid endarterectomy
other adverse events | 7 days
  respiratory complications, such as re-intubation, aspiration Neurologic complication, such as stroke length of hospital stay, ICU admission, length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Aphichat Suphathamwit, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Mutirangura P et al. J Med Assoc Thai 2016; 99 (7): 785-93. 2. Boulanger M et al. Stroke. 2015 Oct;46(10):2843-8. 3. McKee PA et al. N Engl J Med. 1971 Dec 23;285(26):1441-6. 4.Go C et al. Ann Vasc Surg. 2015 Aug;29(6):1265-71. 5.Steinvil A et al. J Am Coll Cardiol. 2011 Feb 15;57(7):779-83. 6.Hoffmann R et al. Heart. 2005 Nov;91(11):1438-41. 7.Sposato LA et al. Journal of the Neurological Sciences. 2011 Oct 15;309(1-2):5-8. 8.Aboyans V et al. Eur Heart J. 2018 Mar 1;39(9):763-816. 9.Varon J, Marik PE. Vasc Health Risk Manag. 2008 Jun; 4(3): 615-627. 10.Landesberg G et al. Circulation. 2009;119:2936-2944